CLINICAL TRIAL: NCT03578900
Title: Quality of Life in a Portuguese Population With Primary Sjögren Syndrome
Brief Title: Quality of Life and Sjögren Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo de Investigação em Bioquímica e Biologia Oral (Other)
Collaborators: University of Lisbon (Other); Portuguese Institute of Rheumatology (Unknown); Dentaid SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: QL2015
Record Dates: First submitted 2018-05-18; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Xerostomia; Hyposalivation; Quality of Life; Sjogren's Syndrome
Keywords: Xerostomia; Hyposalivation; Quality of Life; Sjogren's Syndrome
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome | interventions — Xeros mouthwash

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Xeros Group - Lozenge (Experimental): Application of Xeros system for 15 days. Lozenge (Malic acid 28.56 mg, Xylitol 421,98 mg, Sodium fluoride 0.55 mg) or Spray (Malic acid 1%, Xylitol 10%, Sodium fluoride 0.05%) 4 times a day. Effects on Xerostomia and Quality of Life were determined before and after application by answering the questionnaires.
  Effects of lozenge on hyposalivation and pH variation determined by saliva collection with pre-weighed falcon and a ph electrode at predetermined times during a 20 minute period.
  Interventions: Drug: Xeros
- Mouthwash group (Active Comparator): Application of citric acid based Mouthwash (0,33% citric acid) for 15 days four times a day. Effects on Xerostomia and Quality of Life were determined before and after application by answering the questionnaires.
  Effects of mouthwash on hyposalivation and pH variation determined by saliva collection with pre-weighed falcon and a pH electrode at predetermined times during a 20 minute period.
  Interventions: Drug: Citric Acid based Mouthwash
- Xeros Group - Mouthwash (Experimental): Application of Xeros system for 15 days. Mouthwash (Betaine 1.33%, Xylitol 3.30%, Sodium fluoride 0.05%, Allantoin 0.10%) 2 times a day.
  Effects on Xerostomia and Quality of Life were determined before and after application by answering the questionnaires.
  Interventions: Drug: Xeros
- Xeros Group - Gel (Experimental): Application of Xeros system for 15 days. Gel (Betaine 1%, Aloe Vera 0.05%, Xylitol 10%, Sodium Fluoride 0.0033%) before bed.
  Effects on Xerostomia and Quality of Life were determined before and after application by answering the questionnaires.
  Interventions: Drug: Xeros
- Xeros Group - Toothpaste (Experimental): Application of Xeros system for 15 days. Toothpaste (Betaine 4%, Xylitol 10%, Sodium Fluoride 0.33%, Allantoin 0.10%) 3 times a day.
  Effects on Xerostomia and Quality of Life were determined before and after application by answering the questionnaires.
  Interventions: Drug: Xeros

INTERVENTIONS:
Drug: Xeros
  Arms: Xeros Group - Gel; Xeros Group - Lozenge; Xeros Group - Mouthwash; Xeros Group - Toothpaste
Drug: Citric Acid based Mouthwash
  Arms: Mouthwash group

SUMMARY:
The aims of this study are: To compare salivary pH changes and stimulation efficacy of two different Gustatory Stimulants of Salivation (GSSS) in patients with Primary Sjögren Syndrome (PSS); To evaluate Primary Sjögren syndrome (PSS) impact and gustatory stimulants of salivary secretion (GSSS) on oral health related quality of life measured by a Portuguese version of Oral Health Impact Profile-14 (OHIP-14) and specific Xerostomia assessment questionnaires.

The Products to be used are the Xeros® Dentaid system and a citric based mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* unstimulated whole saliva secretion rate < 0.1 ml/min
* stimulated whole saliva secretion rate > 0.2 ml/min
* above 18 years of age
* Primary Sjogren Syndrome diagnostic according to the European-American Consensus Group

Exclusion Criteria:

* wearer of complete dental prosthesis
* those who were pregnant or lactating
* non-speakers of Portuguese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Time of GSSS induced pH drop below 4.5 | 20 minutes
  On the day that the system is attributed the subject is asked to use one of the products and saliva is collected. pH variation is determined at fixed intervals during 20 minutes. Time in which salivary pH is below 4.5 is calculated as well as the number needed to treat and the absolute risk reduction.
Overall and sub domains scores for each questionnaire | 15 days
  Before and after usage of both products at home, the Summated Xerostomia Inventory-5 (range 0 to 15) to measure subjective feeling of dry mouth, Oral Health Impact Profile-14 (range 0 to 56) to measure quality of life perception related to the oral cavity. This last questionnaire is further divided into 7 subdomains: functional limitation, physical pain, psychological discomfort, physical disability, psychologic disability, social disability and handicap each ranging from 0 to 14.
  In both questionnaires the total score is the result of the sum of the individual scores in each question.
  In both questionnaires the higher the score the worse the outcome. The before and after scores obtained are then compared.

SECONDARY OUTCOMES:
Salivary stimulant induced salivary flow | 20 minutes
  While using one of the two products saliva is collected, weighed and salivary flow is determined at fixed times during 20 minutes.